CLINICAL TRIAL: NCT03691909
Title: A Phase 1/2a Clinical Trial to Assess Safety of a Single IV Infusion of Autologous Adipose-derived Mesenchymal Stem Cells in Adults With Active Rheumatoid Arthritis
Brief Title: Phase 1/2a Clinical Trial to Assess the Safety of HB-adMSCs for the Treatment of Rheumatoid Arthritis
Acronym: HB-adMSCs
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hope Biosciences LLC (Industry)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBRA01
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: arthritis; stem cells; MSCs; adipose MSCs
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Intervention Model Description: A single IV infusion of autologous adipose-derived mesenchymal stem cells (HB-adMSCs) in subjects with clinical diagnosis of RA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Single IV administration of autologous adipose-derived mesenchymal stem cells Baseline laboratory data will be collected prior to infusion; follow up data will be compared against baseline at 1, 3, 6 and 12 months. Joint Assessment 68 will be administered at 1, 3, 6 and 12 months.
  Interventions: Biological: HB-adMSCs

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences autologous adipose-derived mesenchymal stem cells

SUMMARY:
Hope Biosciences is conducting a research study of an investigational product called Hope Biosciences autologous adipose-derived mesenchymal stem cells (abbreviated as HB-adMSCs) as a possible treatment for Rheumatoid Arthritis (RA). The study purpose is to evaluate the safety profile of a single IV infusion of HB-adMSCs in subjects with clinical diagnosis of RA.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, single-dose study in subjects with active Rheumatoid Arthritis (RA). 12-15 patients will be enrolled for the study. The overall objective of this study is to evaluate the safety profile of a single IV infusion of autologous adipose-derived mesenchymal stem cells (HB-adMSCs) in subjects with clinical diagnosis of RA. The primary endpoint of this study is to measure the number and frequency of adverse event(s) and/or severe adverse event(s) throughout the study duration. The second endpoint of this study is to evaluate the ability of HB-adMSCs to alter RA-related inflammation via measuring levels of Tumor Necrosis Factor alpha (TNF-a), Interleukin-6 (IL-6), C-Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR) and Joint Count 66/68 after a single infusion of autologous HB-adMSCs for up to 12-month post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between the ages of 18 and 65
* Patients have active RA as confirmed by the following criteria:

  * ≥ 6 swollen joints and ≥ 6 tender joints at screening (68-joint count)
  * Abnormal CRP result OR abnormal ESR result at screening. Abnormal CRP result at screening OR abnormal ESR defined as:
  * CRP > 4.9 mg/L or ESR > 10mm/hr for men, > 20mm/hr for women
* Patients without current established treatment, or if being treated, patients who are on a stable dose of RA therapy regimen for ≥ 4 weeks prior to screening

Exclusion Criteria:

* Inability to understand and provide signed informed consent

  * Pregnancy, lactation, or, if female of childbearing potential, positive serum β-hCG at screening.
  * Currently diagnosed any malignant neoplasm. Any patient who was successfully treated for cancer and has been disease-free, with no recurrence, for at least 5 years, will be considered.
  * Uncontrolled systemic illness, including, but not limited to: hypertension (systolic >150 mm Hg or diastolic >95 mm Hg); diabetes; renal, hepatic, or cardiac failure or any laboratory abnormality that poses a safety risk to the subject such as:

    * Hemoglobin ≤8.5 g/dL
    * White blood cells (WBCs) ≤3,500/mm3 (3.5 G/L)
    * Any other illness which, in the opinion of the investigator, characterizes the subject as not being a good candidate for the study
  * Participation in another study with an investigational drug or device within 4 weeks prior to treatment or 5 half-lives of the investigational product used (whichever is longer).
  * Positive results of hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCV Ab), and/or human immunodeficiency virus antibody (HIV Ab) tests at screening (excluding patients who are tested positive for HBsAb alone due to a hepatitis B vaccination).
  * Positive history of Treponema pallidum.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Waller, MD, Principal Investigator — Accurate Clinical Research
Locations (1):
- Accurate Clinical Research, Pasadena, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vij R, Stebbings KA, Kim H, Park H, Chang D. Safety and efficacy of autologous, adipose-derived mesenchymal stem cells in patients with rheumatoid arthritis: a phase I/IIa, open-label, non-randomized pilot trial. Stem Cell Res Ther. 2022 Mar 3;13(1):88. doi: 10.1186/s13287-022-02763-w. PMID 35241141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral and 6 participants were recruited through clinicaltrials.gov. First participant was enrolled on 09/25/2018 and last participant was enrolled on 05/23/2019.
Pre-assignment Details: Of 23 screened participants, 15 met inclusion criteria, were enrolled, and given treatment.
Groups:
- Treatment Arm: Single IV administration of Hope Biosciences autologous adipose-derived mesenchymal stem cells (HB-adMSCs).
Period: Overall Study
Arm/Group | Treatment Arm
Started | 15
Per Protocol Population Day 1 | 15
Per Protocol Population Week 1 | 15
Per Protocol Population Week 4 | 14
Per Protocol Population Week 8 | 13
Per Protocol Population Week 12 | 15
Per Protocol Population Week 26 | 14
Per Protocol Population Week 52 | 13
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Single IV administration of Hope Biosciences autologous adipose-derived mesenchymal stem cells (HB-adMSCs) cells.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [38 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Baseline Tumor Necrosis Factor alpha (TNF-a) in patients with acute RA [Median (Inter-Quartile Range); unit: pg/mL] | 1.45 [0.88 to 3.23]
Baseline Interleukin-6 (IL-6) in patients with acute RA [Median (Inter-Quartile Range); unit: pg/mL] | 4.90 [2.90 to 12.1]
Baseline C-Reactive Protein (CRP) in patients with acute RA [Median (Inter-Quartile Range); unit: mg/L] | 10.0 [4.5 to 18.1]
Baseline Erythrocyte Sedimentation Rate (ESR) in patients with acute RA [Median (Inter-Quartile Range); unit: mm/hr] | 43.0 [33.0 to 55.0]
Baseline joint count in patients with acute RA. [Median (Inter-Quartile Range); unit: number of joints]
  Tender | 20.0 [11.0 to 36.0]
  Swollen | 12.0 [8.00 to 19.0]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Adverse Events and Serious Adverse Events
Description: Total number of Adverse Events and Serious Adverse Events across all subjects over 12 months.
Time Frame: 12 months
Population: All participants who received treatment and completed at least 5 of 7 follow up assessments.
Measure: Number; unit: count of events
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
count of events
  Total Adverse Events | 27
  Mild Adverse Events | 15
  Moderate Adverse Events | 8
  Severe Adverse Events | 4
  Treatment Related Mild Adverse Events | 4
  Treatment Related Moderate Adverse Events | 0
  Treatment Related Severe Adverse Events | 0

2. Secondary Outcome: The Effect of Single Injection of HB-adMSCs on TNF-a in Patients With Acute RA
Description: Efficacy is a secondary endpoint for this study and will be assessed by comparing the levels of Tumor Necrosis factor (TNF-a) (pg/mL) measured during trial.
Time Frame: 12 months
Population: All participants who received treatment and completed at least 5 of 7 follow up assessments.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
pg/mL | 1.15 [0.73 to 2.28]
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; p = 0.743, Wilcoxon-signed rank test; Effect Size: 0.09

3. Secondary Outcome: The Effect of Single Injection of HB-adMSCs on IL-6 in Patients With Acute RA
Description: Efficacy is a secondary endpoint for this study and will be assessed by comparing the levels of interleukin 6 (IL-6) (pg/mL) during the trial
Time Frame: 12 months
Population: All participants who received treatment and completed at least 5 of 7 follow up assessments.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
pg/mL | 4.60 [2.75 to 13.9]
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; p = 0.714, Wilcoxon-signed rank test; Effect Size: 0.10

4. Secondary Outcome: The Effect of Single Injection of HB-adMSCs on CRP in Patients With Acute RA
Description: Efficacy is a secondary endpoint for this study and will be assessed by comparing the levels of C-reactive protein (CRP) (mg/L) during the trial
Time Frame: 12 months
Population: All participants who received treatment and completed at least 5 of 7 follow up assessments.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
mg/L | 6.00 [3.00 to 12.0]
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; p = 0.183, Wilcoxon-signed rank test; Effect Size: 0.37

5. Secondary Outcome: The Effect of Single Injection of HB-adMSCs on ESR in Patients With Acute RA
Description: Efficacy is a secondary endpoint for this study and will be assessed by comparing the levels of erythrosedimentation rate (ESR) (mm/hr) during the trial.
Time Frame: 12 months
Population: All participants who received treatment and completed at least 5 of 7 follow up assessments.
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
mm/hr | 34.5 [23.8 to 62.8]
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other; p = 0.775, Wilcoxon-signed rank test; Effect Size: 0.05

6. Secondary Outcome: The Effect of Single Injection of HB-adMSCs on Joint Count in Patients With Acute RA.
Description: Efficacy is a secondary endpoint for this study and will be assessed by comparing the levels of Joint Count 66/68 (# joints - tender and swollen) during the trial.
Time Frame: 12 months
Population: All participants who received treatment and completed at least 5 of 7 follow up assessments.
Measure: Median (Inter-Quartile Range); unit: number of joints
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
number of joints
  Tender | 1.00 [0.00 to 4.00]
  Swollen | 1.00 [0.00 to 3.00]
Statistical Analysis 1: Comparison: Treatment Arm; Tender Joint Count; Test type: Other; p = 0.0008, Wilcoxon-signed rank test; Effect Size: 0.93
Statistical Analysis 2: Comparison: Treatment Arm; Swollen Joint Count; Test type: Other; p = 0.003, Wilcoxon-signed rank test; Effect Size: 0.83

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=15)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (3) — Staph Infection
Intestinal Resection (Surgical and medical procedures) | 1 (1) — Bowel Resection
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) — Bowel Blockage
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) — Complicated Urinary Tract Infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=15)
Rheumatoid arthritis (Immune system disorders) | 2 (2) — Rheumatoid Arthritis Flare/Worsening of RA
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1) — Staph Infection
Rash (Skin and subcutaneous tissue disorders) | 1 (2) — Diffuse Rash/Rash on Abdomen
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of Breath
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) — Bowel Blockage
Anemia (Blood and lymphatic system disorders) | 2 (2) — Anemia/Anemia Chronic Disease
Hematuria (Vascular disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2) — Renal Insufficiency
Eye Pruritus (Eye disorders) | 1 (1) — Right Eyelid Pruritis
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Cyst Right Ear
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck Spasm
Tooth Infection (Infections and infestations) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the protocol signature page, the investigator agreed to the following: "I further agree to treat the results of this Study as confidential information and will not submit the results of the Study for publication without prior written authorization from Hope Biosciences. "

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT03691909/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03691909/SAP_003.pdf